CLINICAL TRIAL: NCT06455293
Title: The Efficacy of Psilocybin Therapy for Depression in Parkinson's Disease
Brief Title: Psilocybin Therapy for Depression in Parkinson's Disease
Acronym: PDP2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Joshua Woolley, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Joshua Woolley, MD, PhD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB#20-32641
Record Dates: First submitted 2024-05-30; First posted 2024-06-12 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease; Depression
Keywords: Parkinson Disease; Depression; Psilocybin; Psilocybin therapy; Movement disorder
MeSH Terms: conditions — Parkinson Disease; Depression; Movement Disorders | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: All participants will receive two doses of psilocybin ranging from low ("microdose") to high. All participants will receive three psilocybin preparation sessions, two administration sessions of a single dose of psilocybin within a therapeutic environment (6-8 hours), five integration sessions, and two follow up visits. All drugs will be orally administered during the dosing sessions. The study procedures will follow best practices for administering psilocybin in clinical trials.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
  This trial is testing various doses of psilocybin. Participants, study staff and clinical assessors will be blinded to individual treatment conditions until study close-out. The clinician administered instruments will be administered by different clinical study staff than the facilitators who provide the preparation, psilocybin therapy, and integration sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psilocybin Administration Session 1 (Experimental): Participants will receive one dose of psilocybin ranging from low ("microdose") to high in a monitored setting with preparation sessions before and integration sessions after.
  Interventions: Drug: Psilocybin
- Psilocybin Administration Session 2 (Experimental): Participants will receive one dose of psilocybin ranging from low ("microdose") to high in a monitored setting with preparation sessions before and integration sessions after.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Single dose of psilocybin ranging from low ("microdose") to high delivered orally with psychological support and monitoring
  Other Names: 4-phosphoryloxy- N,N-dimethyltryptamine

SUMMARY:
The purpose of this study is to understand whether people with Parkinson's Disease and depression have improvement in their symptoms after psilocybin therapy.

DETAILED DESCRIPTION:
This is a randomized controlled trial of oral psilocybin therapy for depression in people with Parkinson's disease (PD). The primary goal is to examine efficacy of psilocybin therapy in this patient population. We will enroll 60 people ages 40 to 80 with clinically diagnosed early to moderate stage Parkinson's disease (Hoehn and Yahr Stage 1-3 during an "on" period), who meet criteria for moderate or greater depression severity and meet all other inclusion and exclusion criteria at screening. Participants will complete two drug administration sessions where they will each receive a dose of oral psilocybin ranging from low ("microdose") to high in a medically monitored setting with psychotherapeutic support. Participants will also complete a series of psychotherapy sessions before and after each drug administration session. Clinical assessments, neuroimaging, non-invasive brain stimulation, and peripheral blood draws will be used to quantify changes in depression, other non-motor and motor symptoms of PD, quality of life, and selected neural and blood-based biomarkers at multiple time points. Follow-up will continue to 3 months after the second session. Primary endpoints will evaluate efficacy, safety, and tolerability of study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 80
* Comfortable speaking and writing in English
* Have neurologist-diagnosed idiopathic Parkinson's disease (PD), Hoehn and Yahr stages 1 to 3 during an "on" phase (time when medication/DBS for parkinsonian motor feature, including bradykinesia and rigidity is in effect)
* Currently experiencing depressive symptoms
* Able to attend all in-person visits at UCSF as well as virtual visits
* Have a primary care provider, neurologist, or psychiatrist who is actively managing or coordinating

Exclusion Criteria:

* Psychotic symptoms involving loss of insight
* Significant cognitive impairment
* Regular use of medications that may have problematic interactions with psilocybin
* A health condition that makes this study unsafe or unfeasible, determined by study physicians

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of psilocybin for improving depression in people living with Parkinson's disease | Baseline to 30 days after first drug dose
  Changes in depression as measured by the Beck Depression Inventory-2 (BDI-2)

SECONDARY OUTCOMES:
Changes in depression severity | 7 days after first drug dose to 90 days after second drug dose
  Measured by Beck Depression Inventory-2 (BDI-2) scores
Changes in clinician-assessed depression | Baseline to 90 days after second drug dose
  Measured by the Montgomery-Asberg Depression Rating Scale (MADRS)
Changes in anxiety | Baseline to 90 days after second drug dose
  Measured by the Parkinson Anxiety Scale (PAS)
Changes in PD symptom severity | Baseline to 90 days after second drug dose
  Measured by the Movement Disorder Society revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
Changes in Quality of Life | Baseline to 90 days after second drug dose
  Measured by the 36-item Short Form survey (SF-36)
Changes in cognitive performance | Baseline to 90 days after second drug dose
  Measured by a multi-task assessment
Safety and tolerability of psilocybin therapy for depression in people with PD | Baseline to 90 days after second drug dose
  Incidence, severity, and frequency of Adverse Events (AEs) including Treatment-Emergent AEs (TEAEs) and Serious AEs (SAEs)
Changes in clinician-rated psychotic symptoms | Baseline to 90 days after second drug dose
  Measured by the Enhanced Scale for the Assessment of Positive Symptoms for Parkinson's Disease (eSAPS-PD)
Subjective effects of psilocybin | Up to 30 and 60 days after Baseline
  Measured by the 5-Dimensional Altered States of Consciousness Rating Scale (5D-ASC)
Participant-reported acceptability of study procedures | 30 days after second drug dose
  Measured by the study-specific Treatment Satisfaction Questionnaire-Participant (TSQ-P)
Care partner/support person reported distress | Baseline to 90 days after second drug dose
  Measured by the Neuropsychiatric Inventory Questionnaire (NPI-Q)

OTHER OUTCOMES:
Changes in peripheral inflammatory markers (exploratory) | Baseline to 90 days after second drug dose
  Measured by blood-based analysis
Changes in brain structure and function (exploratory) | Baseline to 90 days after second drug dose
  Measured by Magnetic Resonance Imaging (MRI) and Transcranial Magnetic Stimulation (TMS)
Changes in participant reported pain (exploratory) | Baseline to 90 days after second drug dose
  Measured by the King's Parkinson's Disease Pain Scale (KPPS)
Changes in participant reported sleep (exploratory) | Baseline to 90 days after second drug dose
  Measured by the Parkinson's Disease Sleep Scale-2 (PDSS-2)
Changes in sleep parameters, physical activity, body temperature, and heart rate (exploratory) | Baseline to 30 days after first drug dose
  Measured by using passive sensing via a wearable device
Evaluation of treatment expectations (exploratory) | Baseline
  Measured by the Treatment Expectancy questionnaire consisting of 6 questions from the Stanford Expectations of Treatment Scale. Rating point scale is from 1 (Strongly disagree) to 7 (Strongly agree). Higher scores represent greater expectations of treatment benefit.
Evaluation of masking procedures (exploratory) | Up to 30 and 60 days after Baseline
  Measured by the study-specific Masking Questionnaire which includes items to assess perceived treatment assignment. Using a 7-point scale, higher scores represent greater certainty.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Woolley, MD,PhD, Principal Investigator — University of California, San Francisco; Ellen Bradley, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No